CLINICAL TRIAL: NCT00423254
Title: A Phase I Multicenter, Open Label, Clinical Trial of Immune Response, Safety and Tolerability of DNA Vector pPRA-PSM With Synthetic Peptides E-PRA and E-PSM in Subjects With Advance Solid Malignancies
Brief Title: Safety and Immune Response to a Multi-component Immune Based Therapy (MKC1106-PP) for Patients With Advanced Cancer.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mannkind Corporation (Industry)
Responsible Party: Mihail Obrocea/Vice President-Oncology - Medical & Regulatory Affairs, MannKind Corporation
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MKC1106-PP-001
Record Dates: First submitted 2007-01-12; First posted 2007-01-18 (Estimated); Last update posted 2010-08-03 (Estimated); Status verified 2010-08

CONDITIONS: Ovarian; Melanoma; Renal; Prostate; Colorectal; Endometrial Carcinoma; Cervical Carcinoma; Testicular Cancer; Thyroid Cancer; Small Cell Lung Carcinoma; Mesothelioma; Breast Carcinoma; Esophageal Carcinoma; Gastric Cancer; Pancreatic Carcinoma; Neuroendocrine Cancer; Liver Cancer; Gallbladder Cancer; Biliary Tract Cancer; Anal Carcinoma; Bone Sarcomas; Soft Tissue Sarcomas; Carcinoma of Unknown Origin, Primary
Keywords: Cancer Vaccine
MeSH Terms: conditions — Melanoma; Endometrial Neoplasms; Uterine Cervical Neoplasms; Testicular Neoplasms; Thyroid Neoplasms; Small Cell Lung Carcinoma; Mesothelioma; Breast Neoplasms; Esophageal Neoplasms; Stomach Neoplasms; Pancreatic Neoplasms; Carcinoma, Neuroendocrine; Liver Neoplasms; Gallbladder Neoplasms; Biliary Tract Neoplasms; Anus Neoplasms; Bone Neoplasms; Sarcoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low Dose Cohort (Experimental)
  Interventions: Biological: PSMA/PRAME
- High Dose Cohort (Experimental)
  Interventions: Biological: PSMA/PRAME

INTERVENTIONS:
Biological: PSMA/PRAME — Low dose
  Arms: Low Dose Cohort
Biological: PSMA/PRAME — high dose
  Arms: High Dose Cohort

SUMMARY:
The present clinical trial is a dose comparison of a multi-component active immunotherapy designed to stimulate an immune reaction to specific tumor associated antigens which are highly expressed on a large number of solid cancers.

DETAILED DESCRIPTION:
The majority of tumors are ignored by the immune system and it was thought for a long time that tumor antigens did not exist. However, recently a number of tumor antigens have been described. These antigens reside on cancer cells and can be recognized by specific T-cells which can ultimately attack and destroy the tumor.

ELIGIBILITY:
Inclusion Criteria:

18 years of age or older Advanced, refractory solid malignancy that is histologically proven Measurable disease ECOG performance status of 0, 1 or 2 Adequate bone marrow reserve as evidenced by a Absolute neutrophil count (ANC) = 1,500/microL; Platelet count = 100,000/microL Adequate renal and hepatic function as evidenced by a serum creatinine = 1.5 mg/dL; Serum total bilirubin = 2.0 mg/dL; Alkaline phosphatase = 3X the ULN for the reference lab (= 5 the ULN for the reference lab for subjects with known hepatic metastases); SGOT/SGPT = 3X the ULN for the reference lab (= 5 the ULN for the reference lab for subjects with known hepatic metastases)

Exclusion Criteria:

Symptomatic central nervous system (CNS) metastases Any autoimmune disorder Positive HIV, hepatitis B or hepatitis C antibody test Any allogeneic transplant Congestive heart failure Affected inguinal lymph nodes (metastatic process) or lack inguinal lymph nodes (resection)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2007-02; Primary Completion 2009-09 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
To determine the immunologic response to the treatment with MKC1106-PP regimen and 2) to determine the safety and adverse event profile of MKC1106-PP | Every 6 Weeks

SECONDARY OUTCOMES:
to determine the blood plasmid levels by PCR analysis | Every 6 Weeks
measure cytokine levels | Every 6 Weeks
to describe any objective tumor responses to the treatment with MKC1106-PP | Every 6 Weeks

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Arizona Cancer Center, Tuscon, Arizona
  - Lombardi Comprehensive Cancer Center at Georgetown, Washington D.C., District of Columbia
  - H Lee Moffitt Cancer Center University of So Florida, Tampa, Florida
  - Nevada Cancer Institute, Sparks, Nevada
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire